CLINICAL TRIAL: NCT02255175
Title: Effects of Estradiol on Neural Reward System and Depression in the Perimenopause
Brief Title: Perimenopausal Effects of Estradiol on Reward Responsiveness
Acronym: PEERS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 13-3572; K12HD001441-15 (NIH); K23MH105569-01A1 (NIH)
Record Dates: First submitted 2014-09-29; First posted 2014-10-02 (Estimated); Results first posted 2019-11-12 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2018-11

CONDITIONS: Perimenopausal Depression
Keywords: Reproductive Affective Disorder; Depression; Perimenopause; Estrogen; Estradiol treatment; Mood Disorders; Estrogen Replacement Therapy; Sex Steroids; Depressive disorder; Mental Disorders; Estradiol; Hormones; Physiological effects of drugs; Reproductive Control Agents
MeSH Terms: conditions — Depression; Mood Disorders; Depressive Disorder; Mental Disorders | interventions — Estradiol; Progesterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Perimenopausal women, depressed (Experimental): Participants will receive transdermal estradiol (100μg/day) for 3 weeks. Participants will receive an additional week of combined estradiol and micronized progesterone (200 mg/day) at the end of the study to precipitate menstruation.
  Interventions: Drug: Estradiol; Drug: Progesterone
- Perimenopausal women, non-depressed (Active Comparator): Participants will receive transdermal estradiol (100μg/day) for 3 weeks. Participants will receive an additional week of combined estradiol and micronized progesterone (200 mg/day) at the end of the study to precipitate menstruation.
  Interventions: Drug: Estradiol; Drug: Progesterone

INTERVENTIONS:
Drug: Estradiol — Participants will receive transdermal estradiol (100μg/day) for 3 weeks
  Other Names: Transdermal estradiol; Climara
Drug: Progesterone — Participants will receive an additional week of combined estradiol and micronized progesterone (200 mg/day) at the end of the study to precipitate menstruation.
  Other Names: Prometrium; Micronized progesterone

SUMMARY:
Using neuroimaging, the investigator will study the effects of estrogen on mood and brain function in perimenopausal women either with or without depression.

DETAILED DESCRIPTION:
Despite decades of research, affective disorders are prevalent and associated with significant morbidity and mortality. Unraveling the pathophysiology of affective disorders has been uniquely challenging because depressive syndromes are heterogeneous and have diverse etiologies. Thus, past studies aimed at identifying neural and genetic biomarkers that would improve the prediction of susceptibility, course of illness, and treatment response have yielded inconsistent results. The investigator proposes to address this problem by studying perimenopausal major depressive disorder (MDD), a depression subtype with a specific endocrine trigger (i.e., ovarian hormone withdrawal). Evidence supporting ovarian hormone withdrawal as a trigger for affective dysfunction in perimenopausal MDD includes the following: perimenopausal women show a temporal association between ovarian hormone withdrawal and the onset of mood symptoms; treatment with estrogen reduces mood symptoms; and blinded estradiol withdrawal re-precipitates depression in women with a history of perimenopausal MDD (manuscript in preparation). Focusing on perimenopausal MDD, a more homogeneous subtype with a specific endocrine trigger, will increase the likelihood of identifying meaningful neurobiological markers.One of the most powerful tools for understanding the neural mediators of MDD is brain imaging. Prior research suggests that the frontostriatal reward system is regulated by estradiol and implicated in MDD. However, neural mechanisms of perimenopausal MDD have never been studied. We will assess the neural reward system in perimenopausal women with and without MDD using functional magnetic resonance imaging (fMRI) at baseline and following estradiol treatment. The central hypothesis is that the neural reward system is hypoactive in perimenopausal MDD, and the antidepressant effects of a three-week transdermal estradiol intervention will be mediated by increased activity in the neural reward system, assessed using fMRI. The investigator will test the hypothesis by executing the following aims:

Aim 1: To measure the frontostriatal response to reward in perimenopausal MDD and test the effects of estradiol on neural activation in perimenopausal women. The investigator will use fMRI at baseline and following estradiol treatment in women with and without MDD to probe frontostriatal reward circuitry.

Aim 2: To quantify motivated behavior at baseline and following estradiol administration in perimenopausal women with and without MDD. Motivated behavior will be operationally defined as the response latency to reward versus non-reward during the fMRI reward task.

Aim 3: To measure the psychological correlates of the frontostriatal response to reward in women with perimenopausal MDD at baseline and following estradiol administration. Depressive symptoms will be assessed at baseline and following estradiol administration.

The results will provide critical information about the neuroendocrine pathophysiology of perimenopausal depression and may subsequently contribute to the development of novel pharmacologic interventions.

ELIGIBILITY:
Inclusion Criteria:

1. Perimenopause Status: We will employ the Stages of Reproductive Aging Workshop (STRAW) criteria70 to confirm perimenopausal status. The stages are primarily based on the characteristics of the menstrual cycle and secondarily on follicle stimulating hormone (FSH) levels. The anchor for the staging system is the final menstrual period (FMP). We will enroll women who have ≥ 2 skipped cycles and an interval of amenorrhea ≥ 60 days, consistent with the late menopause transition (stage -1), and who demonstrate an FSH level > 25 IU/mL. Because extremes of body weight (BMI < 18 or > 30 kg/m2) or a history of chronic menstrual cycle irregularity can contribute to inaccurate reproductive staging, these will serve as additional exclusion criteria;
2. MDD Group Eligibility Criterion: current diagnosis of MDD with an onset associated with menstrual cycle irregularity, and no history of psychiatric illness during the 2 years before the onset of the current depressive episode as determined by the Structured Clinical Interview for DSM-IV-TR (Diagnostic and Statistical Manual-4-Text Revision) for Axis I Disorders (SCID);
3. Control Group Eligibility Criterion: absence of any past or present psychiatric disorder as assessed by the SCID.

Exclusion Criteria:

Patients will not be permitted to enter this protocol if they have any of the following:

1. current medication use (i.e., psychotropics, anti-hypertensives, statins, hormonal preparations, or frequent use of anti-inflammatory agents (> 10 times/month)). Women will be allowed to enroll who take medications without known mood effects (e.g. stable thyroid hormone replacement and occasional (< 5 times/month) use of Ambien)*;
2. pregnant, breastfeeding or trying to conceive;
3. FMP more than 12 months prior to enrollment;
4. history of undiagnosed vaginal bleeding;
5. undiagnosed enlargement of the ovaries;
6. polycystic ovary syndrome;
7. history of breast or ovarian cancer;
8. first degree relative with ovarian cancer;
9. first degree relative with premenopausal onset or bilateral breast cancer;
10. 2+ first degree relatives with breast cancer (regardless of onset);
11. 3+ relatives with postmenopausal breast cancer;
12. abnormal finding in a provider breast exam and/or mammogram;
13. known carrier of BRCA1 or 2 mutation;
14. endometriosis;
15. blood clots in the legs or lungs;
16. porphyria;
17. diabetes mellitus;
18. malignant melanoma;
19. Hodgkin's disease;
20. recurrent migraine headaches that are preceded by aura;
21. gallbladder or pancreatic disease**;
22. heart or kidney disease**;
23. liver disease;
24. cerebrovascular disease (stroke);
25. first degree relative with history of heart attack or stroke;
26. current cigarette smoking;
27. current suicidal ideation or psychosis;
28. past suicide attempts or psychotic episodes requiring hospitalization;
29. chronic depression (i.e., episode(s) lasting 3+ years);
30. recurrent depression (i.e., more than 1 prior episode, not including episodes with postpartum onset)
31. depressive episode(s) within 2 years of enrollment;
32. self-reported claustrophobia
33. peanut allergy

    * all reported prescription medications will be reviewed and cleared by a study physician prior to a participant's enrollment; **participants will be given the opportunity to describe these conditions in the online screening survey. Reported conditions that are acute in nature and/or benign will be reviewed by a study physician and exclusions will be decided case-by-case. All chronic conditions will be exclusionary.

Ages: 44 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2015-10-01; Primary Completion 2018-10-17 (Actual); Study Completion 2018-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Crystal Schiller, PhD, Principal Investigator — University of North Carolina at Chapel Hill Psychiatry Department
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment process included, social media advertising using Facebook, Instagram, and Craigslist; mass emailing using university wide emails and a database of select University of North Carolina (UNC) healthcare patients (Carolina data warehouse); and flyer advertisements placed in university buildings and local businesses.
Pre-assignment Details: Enrolled participants were excluded prior to the start of study intervention due to: exclusionary psychiatric history (i.e. substance abuse, past hypomania, persistent depression), exclusionary gynecological history (i.e. fibroids, abnormal pap), exclusionary medical history (i.e. abnormal lab values), exclusionary medication, and imaging concerns.
Period: Overall Study
Arm/Group | Perimenopausal Women, Depressed | Perimenopausal Women, Non-depressed
Started | 33 | 31
Completed | 16 | 19
Not Completed | 17 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Perimenopausal Women, Depressed | Perimenopausal Women, Non-depressed | Total
Number analyzed (Participants) | 33 | 31 | 64
Age, Continuous [Mean (Full Range); unit: years]
  Age | 50.13 [44 to 55] | 50.76 [44 to 55] | 50.44 [44 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 31 | 64
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White or Caucasion | 23 | 30 | 53
  Race/Ethnicity: Black or African American | 8 | 1 | 9
  Race/Ethnicity: Multi-Racial | 1 | 0 | 1
  Race/Ethnicity: Cuban or Carribean | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Caudate Signal Intensity in Response to Reward During the MID fMRI Task at Pre-treatment
Description: Caudate reactivity to reward during the Monetary Incentive Delay (MID) task was measured between the two groups. During MID the task, participants respond to "win" trials by pressing a button on a button box in the MRI as quickly as possible when the see a target. Reactivity is measured by examining participant's change in blood-oxygen-level dependent (BOLD) (i.e., measurement of oxygen level that is carried to neurons by red blood cells since areas of the brain that are thought to be more "active" or involved in certain tasks require more oxygen) in response to a stimulus of interest (win trials) versus non-stimulus (non-win trials). Percent signal change in BOLD activation between monetary reward versus non-reward is the outcome of interest. Percent signal change is then compared between the two groups at pre-treatment.
Time Frame: Pre-treatment (visit 3)
Measure: Mean (Standard Deviation); unit: percent signal change
Arm/Group | Perimenopausal Women, Depressed | Perimenopausal Women, Non-depressed
Number analyzed (Participants) | 16 | 19
percent signal change | .027 (.105) | .043 (.074)
Statistical Analysis 1: Comparison: Perimenopausal Women, Depressed vs Perimenopausal Women, Non-depressed; Test type: Superiority; p = .620, t-test, 2 sided; t=.501, df=33

2. Primary Outcome: Nucleus Accumbens (NAcc) Signal Intensity in Response to Reward During the MID fMRI Task at Pre-treatment
Description: Nucleus Accumbens (NAcc) reactivity to reward during the Monetary Incentive Delay (MID) task was measured between the two groups. During MID the task, participants respond to "win" trials by pressing a button on a button box in the MRI as quickly as possible when the see a target. Reactivity is measured by examining participant's change in blood-oxygen-level dependent (BOLD) (i.e., measurement of oxygen level that is carried to neurons by red blood cells since areas of the brain that are thought to be more "active" or involved in certain tasks require more oxygen) in response to a stimulus of interest (win trials) versus non-stimulus (non-win trials). Percent signal change in BOLD activation between monetary reward versus non-reward is the outcome of interest. Percent signal change is then compared between the two groups at pre-treatment.
Time Frame: Pre-treatment (visit 3)
Measure: Mean (Standard Deviation); unit: percent signal change
Arm/Group | Perimenopausal Women, Depressed | Perimenopausal Women, Non-depressed
Number analyzed (Participants) | 16 | 19
percent signal change | .045 (.117) | .052 (.108)
Statistical Analysis 1: Comparison: Perimenopausal Women, Depressed vs Perimenopausal Women, Non-depressed; Test type: Superiority; p = .855, t-test, 2 sided; t=.185, df=33

3. Primary Outcome: Putamen Signal Intensity in Response to Reward During the MID fMRI Task at Pre-treatment
Description: Putamen reactivity to reward during the Monetary Incentive Delay (MID) task was measured between the two groups. During MID the task, participants respond to "win" trials by pressing a button on a button box in the MRI as quickly as possible when the see a target. Reactivity is measured by examining participant's change in blood-oxygen-level dependent (BOLD) (i.e., measurement of oxygen level that is carried to neurons by red blood cells since areas of the brain that are thought to be more "active" or involved in certain tasks require more oxygen) in response to a stimulus of interest (win trials) versus non-stimulus (non-win trials). Percent signal change in BOLD activation between monetary reward versus non-reward is the outcome of interest. Percent signal change is then compared between the two groups at pre-treatment.
Time Frame: Pre-treatment (visit 3)
Measure: Mean (Standard Deviation); unit: percent signal change
Arm/Group | Perimenopausal Women, Depressed | Perimenopausal Women, Non-depressed
Number analyzed (Participants) | 16 | 19
percent signal change | .015 (.103) | .004 (.093)
Statistical Analysis 1: Comparison: Perimenopausal Women, Depressed vs Perimenopausal Women, Non-depressed; Test type: Superiority; p = .758, t-test, 2 sided; t=-.310, df=33

4. Primary Outcome: Caudate Signal Intensity in Response to Reward During the MID fMRI Task Following Estradiol Treatment.
Description: Caudate reactivity to reward during the Monetary Incentive Delay (MID) task was measured between the two groups. During MID the task, participants respond to "win" trials by pressing a button on a button box in the MRI as quickly as possible when the see a target. Reactivity is measured by examining participant's change in blood-oxygen-level dependent (BOLD) (i.e., measurement of oxygen level that is carried to neurons by red blood cells since areas of the brain that are thought to be more "active" or involved in certain tasks require more oxygen) in response to a stimulus of interest (win trials) versus non-stimulus (non-win trials). Percent signal change in BOLD activation between monetary reward versus non-reward is the outcome of interest. Percent signal change is then compared between the two groups following treatment.
Time Frame: Post-treatment (visit 6)
Measure: Mean (Standard Deviation); unit: percent signal change
Arm/Group | Perimenopausal Women, Depressed | Perimenopausal Women, Non-depressed
Number analyzed (Participants) | 16 | 19
percent signal change | .005 (.079) | .026 (.103)
Statistical Analysis 1: Comparison: Perimenopausal Women, Depressed vs Perimenopausal Women, Non-depressed; Test type: Superiority; p = .518, t-test, 2 sided; t=.653, df=33

5. Primary Outcome: Nucleus Accumbens (NAcc) Signal Intensity in Response to Reward During the MID fMRI Task Following Estradiol Treatment.
Description: Nucleus accumbens (NAcc) reactivity to reward during the Monetary Incentive Delay (MID) task was measured between the two groups. During MID the task, participants respond to "win" trials by pressing a button on a button box in the MRI as quickly as possible when the see a target. Reactivity is measured by examining participant's change in blood-oxygen-level dependent (BOLD) (i.e., measurement of oxygen level that is carried to neurons by red blood cells since areas of the brain that are thought to be more "active" or involved in certain tasks require more oxygen) in response to a stimulus of interest (win trials) versus non-stimulus (non-win trials). Percent signal change in BOLD activation between monetary reward versus non-reward is the outcome of interest. Percent signal change is then compared between the two groups following treatment.
Time Frame: Post-treatment (visit 6)
Measure: Mean (Standard Deviation); unit: percent signal change
Arm/Group | Perimenopausal Women, Depressed | Perimenopausal Women, Non-depressed
Number analyzed (Participants) | 16 | 19
percent signal change | .040 (.110) | .059 (.118)
Statistical Analysis 1: Comparison: Perimenopausal Women, Depressed vs Perimenopausal Women, Non-depressed; Test type: Superiority; p = .645, t-test, 2 sided; t=.465, df=33

6. Primary Outcome: Putamen Signal Intensity in Response to Reward During the MID fMRI Task Following Estradiol Treatment.
Description: Putamen reactivity to reward during the Monetary Incentive Delay (MID) task was measured between the two groups. During MID the task, participants respond to "win" trials by pressing a button on a button box in the MRI as quickly as possible when the see a target. Reactivity is measured by examining participant's change in blood-oxygen-level dependent (BOLD) (i.e., measurement of oxygen level that is carried to neurons by red blood cells since areas of the brain that are thought to be more "active" or involved in certain tasks require more oxygen) in response to a stimulus of interest (win trials) versus non-stimulus (non-win trials). Percent signal change in BOLD activation between monetary reward versus non-reward is the outcome of interest. Percent signal change is then compared between the two groups following treatment.
Time Frame: Post-treatment (visit 6)
Measure: Mean (Standard Deviation); unit: percent signal change
Arm/Group | Perimenopausal Women, Depressed | Perimenopausal Women, Non-depressed
Number analyzed (Participants) | 16 | 19
percent signal change | -.030 (.068) | .032 (.073)
Statistical Analysis 1: Comparison: Perimenopausal Women, Depressed vs Perimenopausal Women, Non-depressed; Test type: Superiority; p = .015, t-test, 2 sided; t=2.56, df=33

7. Secondary Outcome: Response Latency to Reward During the MID fMRI Task at Pre-treatment
Description: Time (ms) between stimulus and response will be measured during the Monetary Incentive Delay (MID) task during the win trials. During MID the task, participants need to select the correct response during "win" and "lose" conditions by pressing a button on a button box in the MRI.
Time Frame: Pre-treatment (visit 3)
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Perimenopausal Women, Depressed | Perimenopausal Women, Non-depressed
Number analyzed (Participants) | 16 | 19
Milliseconds | 204.17 (25.11) | 209.63 (20.71)
Statistical Analysis 1: Comparison: Perimenopausal Women, Depressed vs Perimenopausal Women, Non-depressed; Test type: Superiority; p = .486, t-test, 2 sided; t=.705, df=33

8. Secondary Outcome: Response Latency to Reward During the MID fMRI Task Following Estradiol Treatment
Description: Time (ms) between stimulus and response will be measured during reward trials of the Monetary Incentive Delay (MID) task. During MID the task, participants need to select the correct response during "win" and "lose" conditions by pressing a button on a button box in the MRI.
Time Frame: Post-treatment (visit 6)
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Perimenopausal Women, Depressed | Perimenopausal Women, Non-depressed
Number analyzed (Participants) | 16 | 19
Milliseconds | 190.68 (34.98) | 193.43 (39.60)
Statistical Analysis 1: Comparison: Perimenopausal Women, Depressed vs Perimenopausal Women, Non-depressed; Test type: Superiority; p = .831, t-test, 2 sided; t=.216, df=33

9. Secondary Outcome: Change in Inventory of Depression and Anxiety Symptoms (IDAS) Dysphoria Scores
Description: The Dysphoria Scale of the Inventory of Depression and Anxiety Symptoms (IDAS) will be used to assess the change in depressive symptom severity. The IDAS Dysphoria Scale consists of 10 items and uses a 5-point Likert-type scale, ranging from 1 to 5 with 1 indicating "not at all" and 5 indicating "extremely". As such, the range of possible scores is 10 to 50. The Dysphoria scale includes items assessing feelings of depression, inadequacy, psychomotor agitation, guilt, discouragement, anhedonia, poor concentration, difficulty with decision-making, psychomotor retardation, and worry. Higher scores indicate worse depression symptoms.
Time Frame: Assessed at pre- and post-treatment (visits 3 and 6)
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Perimenopausal Women, Depressed, Baseline; Perimenopausal Women, Non-depressed, Baseline; Perimenopausal Women, Depressed, Following Estradiol Treatment; Perimenopausal Women, Non-depressed, Following Estradiol: Participants will receive transdermal estradiol (100μg/day) for 3 weeks. Participants will receive an additional week of combined estradiol and micronized progesterone (200 mg/day) at the end of the study to precipitate menstruation.
  Estradiol: Participants will receive transdermal estradiol (100μg/day) for 3 weeks
  Progesterone: Participants will receive an additional week of combined estradiol and micronized progesterone (200 mg/day) at the end of the study to precipitate menstruation.
Arm/Group | Perimenopausal Women, Depressed, Baseline | Perimenopausal Women, Non-depressed, Baseline | Perimenopausal Women, Depressed, Following Estradiol Treatment | Perimenopausal Women, Non-depressed, Following Estradiol
Number analyzed (Participants) | 16 | 19 | 16 | 19
score on a scale | 24.56 (1.47) | 13.79 (1.35) | 15.25 (1.13) | 11.84 (1.04)
Statistical Analysis 1: Comparison: Perimenopausal Women, Depressed, Baseline vs Perimenopausal Women, Non-depressed, Baseline vs Perimenopausal Women, Depressed, Following Estradiol Treatment vs Perimenopausal Women, Non-depressed, Following Estradiol; Test type: Superiority; p = .0002, Repeated measures ANOVA; F(1,33)=17.91

ADVERSE EVENTS:
Time Frame: Adverse event data was tracked over a participants time in the protocol (1 month), all unresolved adverse events were tracked by the investigator until the events were resolved, the subject was lost to follow-up, or the adverse event was otherwise explained.
Arm/Group | Perimenopausal Women, Depressed | Perimenopausal Women, Non-depressed
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/31
Other Adverse Events (participants affected / at risk) | 16/33 | 17/31
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Perimenopausal Women, Depressed (N=33) | Perimenopausal Women, Non-depressed (N=31)
Itchiness at patch site (Skin and subcutaneous tissue disorders) | 5 (5) | 4 (4)
Headaches (Nervous system disorders) | 4 (4) | 4 (4)
Breast Tenderness (Reproductive system and breast disorders) | 6 (6) | 3 (3) — Breast fullness or tenderness.
Cramps (Reproductive system and breast disorders) | 5 (5) | 3 (3) — menstrual type cramps, abdominal pain and tenderness, sensitive groin
Bloating (Endocrine disorders) | 2 (2) | 2 (2) — Water retention or bloating
Nausea (Gastrointestinal disorders) | 3 (3) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2)
Menstrual Bleeding (Reproductive system and breast disorders) | 2 (2) | 2 (2)
Hot Flashes (Endocrine disorders) | 2 (2) | 1 (1)
Waking during the night (General disorders) | 0 (0) | 2 (2)
Acne (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Lower Back Pain (General disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-12): https://cdn.clinicaltrials.gov/large-docs/75/NCT02255175/Prot_SAP_000.pdf